CLINICAL TRIAL: NCT01170611
Title: Prevention of Atrial Arrhythmia in Patients Without AV Conduction Disease
Brief Title: Prevention of Atrial Arrhythmia in Patients Without Atrioventricular (AV) Conduction Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: WIEGAND, Universitätklinik. Lübeck - Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREFACE-IPRE03; IPRE03
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Sinus Node Dysfunction; Brady Tachy Syndrome
MeSH Terms: conditions — Sick Sinus Syndrome

ARMS (1):
- AAISAFER alone - AAISAFER+PREVENTIVE ALGORITHM - DDD (Experimental)
  Interventions: Device: PACEMAKER SYMPHONY 2550

INTERVENTIONS:
Device: PACEMAKER SYMPHONY 2550

SUMMARY:
This clinical investigation is a prospective, single-blinded, randomized trial. The primary objective concerns the safety and effectiveness of the AAIsafeR mode with the preventive algorithms.

DETAILED DESCRIPTION:
In this study, patients are randomized to DDD mode, AAIsafeR mode, or AAIsafeR mode plus atrial arrhythmia preventive algorithms. The atrial arrhythmia (AA) burden serves as the primary measure of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* A pacemaker indication for sinus node dysfunction and/or brady-tachy syndrome OR already implanted for less than three months for the mentioned reasons and supplied with a symphony 2550 DR at time of inclusion AND
* A PR interval <250ms AND
* Documented atrial arrhythmia in the past year
* Medication for anti-arrhythmic must be stable for at least one month (2 months for amiodarone) prior to enrollment
* Patients must have less than two known cardioversions within the last year
* Patient has signed a consent form after having received the appropriate information

Exclusion Criteria:

* Need a replacement pacemaker device
* Have an unknown PR interval
* Known AV block ≥ 250 ms PR interval
* Minor and/or pregnant woman
* Patients enrolled in other clinical trials
* Patients with sustained ventricular arrhythmia
* Patients with severe coronary artery disease (at the discretion of the investigator)
* Patients with advanced cardiomyopathy (at the discretion of the investigator)
* Patients who have sustained a myocardial infarction or undergone cardiac surgery within the past 30 days
* Patients with unstable angina pectoris
* Patients whose life expectancy is less than 1 year
* Patients who are unlikely to return for required follow-up visits
* Patients who present with permanent atrial arrhythmia or those who usually require cardioversion to terminate such arrhythmia and/or
* Patients whose physician plans to add or change medical treatment because of AA episodes during the follow-up period.
* Patient unable to understand the purpose of the study or refusing to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Atrial arrhythmia burden

CONTACTS AND LOCATIONS:
Locations (52):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Baywood Heart Hospital, Mesa, Arizona
  - Brentwood Biomedical Research Institute, Los Angeles, California
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Passaic Beth Israel Regional Medical Center, Passaic, New Jersey
  - NorthEast Medical Center, Concord, North Carolina
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Lancaster Regional Medical Center, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
- Belgium (8):
  - OLV Aalst, Aalst
  - Cliniques Sud Luxembourg, Arlon
  - Clinique Saint-Jean, Brussels
  - Algemeen Ziekenhuis Sint-Dimpna, Geel
  - Centre Hospitalier Hutois, Huy
  - CHU Tivoli, La Louvière
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
  - UCL Mont-Godinne, Yvoir
- France (21):
  - CHG d'Albi, Albi
  - CHRU du Morvan Hôpital la Cavale Blanche, Brest
  - Hospice St-Jacques-Hôpital G.Montpied, Clermond-Ferrand
  - Hôpital Henri Mondor, Créteil
  - C.H.I. du Val d'Ariège, Foix
  - CHRU de Grenoble Hôpital Michallon, Grenoble
  - Polyclinique du Bois, Lille
  - CHU de Limoges Hôpital Dupuytren, Limoges
  - Clinique Clairval, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Polyclinique de Gentilly, Nancy
  - Nouvelles Cliniques Nantaises, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital Pitié-Salpêtrière, Paris
  - InParys CLINIQUE BIZET, Paris
  - CHU Haut l'Evêque, Pessac
  - CHU Pontchaillou, Rennes
  - CHU - Hôpital Charles Nicolle, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - Centre Hospitalier Rangueil, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - Hufeland Krankenhaus GmbH, Bad Langensalza
  - Charite Campus Virchow, Berlin
  - Kliniken der Stadt Köln, Cologne
  - Universitätklinikum Leipzig, Leipzig
  - Universitätklinik. Lübeck, Lübeck
  - Klinikum Lüdenscheid, Lüdenscheid
  - Johannes Gutenberg-Universität - Mainz Klinikum, Mainz
  - Klinikum Memmingen, Memmingen
- Ospedale San Tommaso dei Battuti, Portogruaro, VE, Italy
- CH Princesse Grace, Monaco, Monaco
- Complejo Hospitalario Universitario de Vigo (CHUVI), Pontevedra, Spain
- United Kingdom (2):
  - Eastbourne District General Hospital, Eastbourne, East Sussex
  - St Peters Hospital, Chertsey, Surrey